CLINICAL TRIAL: NCT07369102
Title: Esketamine With or Without Psychedelic Preparation and Integration for Treatment-Resistant Depression: A Randomized Controlled Trial
Brief Title: Esketamine With or Without Integration Therapy for Treatment-Resistant Depression
Acronym: KIND-PR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Paulina Rullan-Farinacci, Principal Investigator, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2507449648
Record Dates: First submitted 2025-08-22; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Treatment-resistant Depression (TRD)
Keywords: esketamine; Treatment-Resistant Depression; Spravato; Ketamine-Assisted Psychotherapy; Psychedelic Integration; Depression; Integration Therapy; Preparation and Integration; Mental Health; Dissociation; Intranasal Esketamine; Randomized Controlled Trial; Psychiatric Treatment; Therapeutic Support; Psychedelic Medicine
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Psychological Well-Being; Dissociative Disorders | interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel assignment, randomized controlled trial comparing esketamine treatment with and without integration therapy sessions in adults with treatment-resistant depression.
Who Masked: Outcomes Assessor
Masking Description: Independent clinician raters administering primary outcome measures (e.g., MADRS) will be blinded to participant group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esketamine With Integration Therapy (Experimental): Participants in this arm will receive FDA-approved intranasal esketamine (Spravato®) twice weekly during the acute phase (weeks 1-4), followed by weekly or biweekly dosing during the maintenance phase (weeks 5-8), based on clinical response. In addition, participants will receive brief, structured therapeutic sessions for preparation and integration before and after each dosing session. These sessions are designed to support emotional processing, meaning-making, and therapeutic engagement.
  Interventions: Drug: Esketamine hydrochloride (intranasal); Behavioral: Integration Therapy
- Esketamine Without Integration Therapy (Active Comparator): Participants in this arm will receive FDA-approved intranasal esketamine (Spravato®) twice weekly during the acute phase (weeks 1-4), followed by weekly or biweekly dosing during the maintenance phase (weeks 5-8), based on clinical response. No additional psychotherapeutic support will be provided beyond standard clinical monitoring and psychiatric care.
  Interventions: Drug: Esketamine hydrochloride (intranasal)

INTERVENTIONS:
Drug: Esketamine hydrochloride (intranasal) — Intranasal esketamine (Spravato®), administered under medical supervision in accordance with FDA guidelines for treatment-resistant depression. Dosing schedule includes twice-weekly administration during weeks 1-4 (acute phase), followed by weekly or biweekly administration during weeks 5-8 (maintenance phase), based on clinical response and tolerability. All dosing occurs in a clinical setting with standard monitoring for at least two hours post-administration.
  Other Names: Spravato
Behavioral: Integration Therapy — Brief, structured psychotherapeutic sessions delivered before and after each esketamine dose, based on psychedelic-assisted therapy principles. Sessions are designed to support emotional safety, preparation for the treatment experience, and integration of psychological content that may arise. Conducted by trained clinicians following a standardized framework developed for this study. Only participants in the experimental arm receive this intervention.
  Arms: Esketamine With Integration Therapy

SUMMARY:
This study will explore the effects of esketamine (Spravato®), an FDA-approved nasal spray, on adults diagnosed with treatment-resistant depression (TRD). All participants will receive esketamine as prescribed by a healthcare professional in a clinical setting.

The purpose of this research is to understand whether adding therapeutic support in the form of preparation and integration sessions - before and after the esketamine doses - can enhance the treatment experience and lead to longer-lasting improvements in mood and functioning.

Participants will be randomly assigned to one of two groups:

Esketamine with therapeutic support sessions (integration group) Esketamine without additional support (standard care group) Both groups will receive standard monitoring and psychiatric evaluation during the study. The support sessions offered in the integration group are designed to help participants prepare for their treatment sessions and make sense of their experiences afterward, using a structured, evidence-based approach.

The study will last approximately 8 weeks per participant, with follow-up assessments. The goal is to learn whether integration therapy can improve treatment outcomes, safety, and satisfaction for individuals with depression that hasn't responded to other treatments.

DETAILED DESCRIPTION:
This is a single-site, randomized, controlled trial evaluating the effects of therapeutic preparation and integration on the clinical outcomes and subjective experience of intranasal esketamine treatment in adults with treatment-resistant depression (TRD).

All participants will receive FDA-approved intranasal esketamine (Spravato®) twice weekly in accordance with current clinical guidelines. Participants will be randomly assigned to one of two arms:

Integration Arm: Esketamine with brief, structured preparation and integration sessions conducted by a trained clinician Control Arm: Esketamine without additional psychotherapeutic support beyond standard care Therapeutic support in the integration arm is informed by existing psychedelic-assisted therapy frameworks and consists of brief, manualized sessions designed to enhance safety, emotional processing, and meaning-making. These sessions aim to help participants prepare psychologically for their esketamine experiences and to integrate insights or emotional responses afterward.

The primary outcome is change in depression severity, as measured by the Montgomery-Åsberg Depression Rating Scale (MADRS). Secondary outcomes include measures of emotional regulation, therapeutic alliance, treatment acceptability, and dissociative experiences. Exploratory measures will examine participants' engagement with integration, perceived coherence of their experience, and overall satisfaction.

This study seeks to address a current gap in the literature by evaluating the role of structured psychological support in esketamine treatment for depression. While esketamine has demonstrated rapid antidepressant effects, the variability in subjective response and relapse rates suggests that adjunctive support may be beneficial. By including both quantitative and qualitative measures, the study aims to generate data to inform more holistic and patient-centered models of esketamine treatment.

All study procedures will be conducted at a licensed clinical site under the supervision of qualified healthcare professionals. The protocol has received ethical approval from an institutional review board (IRB), and all participants will provide informed consent prior to participation.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults aged 21 to 65 years.
* Diagnosis: Current Major Depressive Disorder (MDD) as confirmed by Structured Clinical Interview for DSM5 (SCID-5).
* Treatment Resistance: Failure to achieve remission with at least two antidepressants of adequate dose and duration (TRD criteria) as confirmed by SCID-5.
* Symptom Severity: Baseline Montgomery-Åsberg Depression Rating Scale (MADRS) ≥30.
* Suicidal Ideation: Participants with baseline passive or active suicidal ideation may be included, provided they do not meet criteria for inpatient admission and are deemed clinically stable for outpatient care. This will be measured with the Columbia Suicide Severity Rating Scale (C-SSRS).
* Consent: Ability to understand and voluntarily provide written informed consent.
* Contraception: For participants of reproductive potential, willingness to use at least one highly effective method of contraception (e.g., intrauterine device, hormonal contraception, sterilization) or two effective methods (e.g., barrier method plus spermicide) during the study and for at least one month after the final esketamine dose. Contraceptive method(s) will be documented at baseline via self-report on a standardized form and reaffirmed at each esketamine session by research staff. Participants who become pregnant or are unable to confirm adequate contraception will be withdrawn from the study for safety reasons.
* Availability: Willingness and ability to attend all scheduled sessions and complete study procedures.
* Motivation for Engagement: Demonstrates willingness and psychological readiness to engage in guided reflective work before and after esketamine dosing (as assessed during clinical intake).

Exclusion Criteria:

* Acute Suicide Risk: Immediate need for inpatient psychiatric hospitalization due to suicidal ideation with plan or intent as identified through the C-SSRS.
* Psychotic or Bipolar Disorders: Current diagnosis of bipolar I disorder (manic phase), schizophrenia, schizoaffective disorder, or other primary psychotic disorders if stated by participants as a past diagnosis or identified during the SCID-5.
* Substance Use Disorder: Active moderate to severe substance use disorder (except nicotine) in the past 6 months as self-identified by participant or during the SCID-5.
* Cognitive/Developmental Impairments: Intellectual disability, dementia, or other cognitive/developmental disorders that impair ability to engage meaningfully in structured psychotherapeutic sessions such as preparation or integration, per clinician judgment.
* Medical Contraindications: Any medical condition judged to pose undue risk during esketamine administration (e.g., aneurysmal vascular disease, arteriovenous malformation, history of intracerebral hemorrhage, or hypersensitivity to esketamine/ketamine).
* Pregnancy/Breastfeeding: Current pregnancy or breastfeeding.
* Ongoing Structured Psychotherapy Likely to Confound Outcomes: Participation in any formal psychotherapy within the past 3 months that involves structured, weekly sessions focused on behavioral change or emotional processing (e.g., CBT, ACT, psychodynamic therapy), unless the therapy was completed or stabilized at a low-intensity level for at least 8 weeks prior to enrollment.
* Prior Non-Response to Esketamine: Six or more prior esketamine (≥56 mg) or IV ketamine sessions (0.4-0.7 mg/kg) without clinical response.
* Recent Ketamine Use: Use of ketamine/esketamine in the past 12 weeks.
* Inability to Consent: Any condition rendering the participant unable to provide informed consent.
* Prior Enrollment: Previous participation in this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Depression Severity as Assessed by MADRS | Baseline and end of acute treatment at 8 weeks
  Change in Montgomery-Åsberg Depression Rating Scale (MADRS) total score from baseline to the end of acute treatment. The MADRS is a clinician-rated scale assessing depressive symptom severity, with scores ranging from 0 to 60. Higher scores indicate more severe depression; lower scores indicate symptom improvement.

SECONDARY OUTCOMES:
Proportion of Participants Achieving Treatment Response (≥50% Reduction in MADRS) | From enrollment (baseline) to the end of acute treatment at 8 weeks
  Number of participants achieving treatment response, defined as a ≥50% reduction in MADRS total score from baseline. MADRS scores range from 0 to 60, with higher scores indicating greater depression severity.
Proportion of Participants Achieving Remission (MADRS <10) | At the end of acute treatment at 8 weeks
  Number of participants achieving remission, defined as a MADRS total score below 10 at the end of acute treatment. MADRS scores range from 0 to 60, with lower scores indicating fewer depressive symptoms.
Proportion of Participants Experiencing Depressive Relapse Confirmed by SCID-5 | From achievement of remission through 6 months after completion of acute treatment
  Number of participants meeting DSM-5 criteria for a new major depressive episode after achieving remission, as assessed using the Structured Clinical Interview for DSM-5 (SCID-5). This is a categorical diagnostic outcome (yes/no).
Change From Baseline in Functional Impairment as Assessed by WSAS | Baseline and end of acute treatment at 8 weeks
  Change in Work and Social Adjustment Scale (WSAS) total score from baseline to the end of acute treatment. WSAS scores range from 0 to 40, with higher scores indicating greater functional impairment and lower scores indicating better functioning.
Change From Baseline in Suicidality as Assessed by C-SSRS | Baseline and end of acute treatment at 8 weeks
  Change in suicidal ideation and behavior severity as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS). The scale includes ordinal severity categories, with higher scores indicating greater suicidality risk.

OTHER OUTCOMES:
Subjective Experience Following Esketamine Administration (Qualitative Reflections) | Within 72 hours after dosing sessions occurring at Weeks 4 and 8
  Subjective experiences assessed through semi-structured interviews and written reflections exploring emotional, perceptual, and psychological experiences following esketamine sessions. Data will be analyzed using thematic qualitative analysis. This outcome does not use a numeric score.
Engagement With Psychedelic Integration as Assessed by Integration Scales | Within 72 hours after each integration session and at the end of acute treatment at 8 weeks
  Engagement with preparation and integration processes assessed using Psychedelic Integration Scales. Scores reflect perceived meaning-making, insight, and behavioral integration. Scale scores range from lowest possible score (minimal engagement) to highest possible score (high engagement and integration); higher scores indicate greater integration.
Treatment Credibility and Expectancy as Assessed by the CEQ | Baseline: after the first preparation session and prior to the first esketamine dosing session
  Treatment credibility and expectancy assessed using the Credibility/Expectancy Questionnaire (CEQ). CEQ items are scored on Likert scales, with higher scores indicating greater perceived credibility and expectancy of benefit.
Therapeutic Alliance as Assessed by the Working Alliance Inventory-Short Form (WAI-SF) | At Week 4 of acute treatment
  Therapeutic alliance assessed using the Working Alliance Inventory-Short Form (WAI-SF), which measures agreement on goals, tasks, and therapeutic bond. Scores range from 12 to 84, with higher scores indicating stronger therapeutic alliance.
Dissociative Symptoms as Assessed by the CADSS | Immediately after each esketamine dosing session during the acute treatment phase
  Dissociative symptoms assessed using the Clinician-Administered Dissociative States Scale (CADSS). Total scores range from 0 to 92, with higher scores indicating greater dissociative symptom severity.
Mystical-Type Experience as Assessed by the MEQ-30 | Within 24 hours after dosing sessions 2 and 4 during the acute treatment phase
  Mystical-type experiences assessed using the Mystical Experience Questionnaire-30 (MEQ-30), including total and subscale scores. Scores range from 0 to 5 per item, with higher scores indicating greater intensity of mystical-type experiences.
Altered States of Consciousness as Assessed by the 5D-ASC | Within 24 hours after dosing sessions 2 and 4 during the acute treatment phase
  Altered states of consciousness assessed using the Five-Dimensional Altered States of Consciousness (5D-ASC) questionnaire. Subscale scores range from 0 to 100, with higher scores indicating greater intensity of altered states.
Change From Baseline in Emotion Regulation Difficulties as Assessed by DERS | Baseline and end of acute treatment at 8 weeks
  Change in Difficulties in Emotion Regulation Scale (DERS) total score from baseline to the end of acute treatment. Total scores range from 36 to 180, with higher scores indicating greater difficulty with emotion regulation.
Patient Satisfaction as Assessed by the Client Satisfaction Questionnaire-8 (CSQ-8) | At the end of acute treatment at 8 weeks and 6 months after completion of acute treatment
  Patient satisfaction assessed using the Client Satisfaction Questionnaire-8 (CSQ-8). Total scores range from 8 to 32, with higher scores indicating greater satisfaction with care.
Negative Treatment Effects as Assessed by the Negative Effects Questionnaire (NEQ) | At the end of acute treatment at 8 weeks and 6 months after completion of acute treatment
  Negative treatment effects assessed using the Negative Effects Questionnaire (NEQ), including total and subscale scores. Higher scores indicate greater perceived negative effects of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Karen G Gonzalez-Martinez, MD, MSc, Study Chair — University of Puerto Rico, Medical Sciences Campus, Department of Psychiatry
Locations (2):
- Puerto Rico (2):
  - Pravan Foundation, San Juan
  - University of Puerto Rico, Department of Psychiatry, San Juan

IPD SHARING:
Plan to Share IPD: Undecided
The investigators may consider sharing de-identified individual participant data upon study completion, subject to IRB approval, institutional policy, and data use agreements.

REFERENCES:
- [Background] Wilkinson ST, Rhee TG, Joormann J, Webler R, Ortiz Lopez M, Kitay B, Fasula M, Elder C, Fenton L, Sanacora G. Cognitive Behavioral Therapy to Sustain the Antidepressant Effects of Ketamine in Treatment-Resistant Depression: A Randomized Clinical Trial. Psychother Psychosom. 2021;90(5):318-327. doi: 10.1159/000517074. Epub 2021 Jun 29. PMID 34186531
- [Background] Dore J, Turnipseed B, Dwyer S, Turnipseed A, Andries J, Ascani G, Monnette C, Huidekoper A, Strauss N, Wolfson P. Ketamine Assisted Psychotherapy (KAP): Patient Demographics, Clinical Data and Outcomes in Three Large Practices Administering Ketamine with Psychotherapy. J Psychoactive Drugs. 2019 Apr-Jun;51(2):189-198. doi: 10.1080/02791072.2019.1587556. Epub 2019 Mar 27. PMID 30917760
- [Background] Gorman I, Nielson EM, Molinar A, Cassidy K, Sabbagh J. Psychedelic Harm Reduction and Integration: A Transtheoretical Model for Clinical Practice. Front Psychol. 2021 Mar 15;12:645246. doi: 10.3389/fpsyg.2021.645246. eCollection 2021. PMID 33796055
- [Background] Aixalà M. Psychedelic Integration: Psychotherapy for Non-Ordinary States of Consciousness. Santa Cruz, CA: MAPS; 2021.
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Background] Popova V, Daly EJ, Trivedi M, Cooper K, Lane R, Lim P, Mazzucco C, Hough D, Thase ME, Shelton RC, Molero P, Vieta E, Bajbouj M, Manji H, Drevets WC, Singh JB. Efficacy and Safety of Flexibly Dosed Esketamine Nasal Spray Combined With a Newly Initiated Oral Antidepressant in Treatment-Resistant Depression: A Randomized Double-Blind Active-Controlled Study. Am J Psychiatry. 2019 Jun 1;176(6):428-438. doi: 10.1176/appi.ajp.2019.19020172. Epub 2019 May 21. PMID 31109201
- [Background] Daly EJ, Trivedi MH, Janik A, Li H, Zhang Y, Li X, Lane R, Lim P, Duca AR, Hough D, Thase ME, Zajecka J, Winokur A, Divacka I, Fagiolini A, Cubala WJ, Bitter I, Blier P, Shelton RC, Molero P, Manji H, Drevets WC, Singh JB. Efficacy of Esketamine Nasal Spray Plus Oral Antidepressant Treatment for Relapse Prevention in Patients With Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Sep 1;76(9):893-903. doi: 10.1001/jamapsychiatry.2019.1189. PMID 31166571
- See also: Institutional Site — https://md.rcm.upr.edu/psychiatry/
- See also: Study Site — https://pravanfoundation.org/en/
- See also: Janssen Pharmaceuticals press release announcing FDA approval of Spravato® (esketamine) for treatment-resistant depression — https://www.jnj.com/media-center/press-releases/spravato-esketamine-approved-in-the-u-s-as-the-first-and-only-monotherapy-for-adults-with-treatment-resistant-depression